CLINICAL TRIAL: NCT05569564
Title: Evaluation of Osseodensification Versus Osseodensification With Ridge Splitting in Horizontally Deficient Ridge (A Randomized Clinical Study)
Brief Title: Evaluation of Osseodensification Versus Osseodensification With Ridge Splitting in Horizontally Deficient Ridge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Farouk Mohamed Hussein Elsobky, Assistant lecturer of periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec ID032211
Record Dates: First submitted 2022-09-29; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Osseodensification
Keywords: Osseodensification; Alveolar ridge splitting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osseodensification with ridge splitting (Experimental): Ridge splitting followed by osseodensification using osseodensifying burs .
  Interventions: Procedure: Ridge splitting followed by ossedensificaion; Procedure: Osseodensification
- Osseodensification (Active Comparator): osseodensification will be performed using osseodensifying burs.
  Interventions: Procedure: Osseodensification

INTERVENTIONS:
Procedure: Ridge splitting followed by ossedensificaion — Ridge splitting followed by ossedensificaion with osseodensifying burs.
  Arms: Osseodensification with ridge splitting
Procedure: Osseodensification — Pilot drill is used to make the initial osteotomy to the desired depth, then osseodensifying burs will be used in sequence, gradually wider diameter in a counterclockwise rotation and bouncing motion under profuse saline irrigation

SUMMARY:
Osseodensification is a method of biomechanical bone preparation where specially designed burs increase density of bone as they expand an osteotomy. These osseodensifying burs combine advantages of osteotome bone preservation with the standard traditional drilling burs speed and tactile control. The investigators compared ridge splitting followed by osseodensification versus osseodensification in terms of buccolingual ridge expansion both clinically and radiographically.

DETAILED DESCRIPTION:
Sixteen patients will be randomly allocated into two groups. Ridge splitting followed by osseodensification will be performed with simultaneous implant placement in group I.

Osseodensification will be performed with simultaneous implant placement in group II.

Alveolar ridge width and Implant stability will be assessed clinically. Alveolar ridge width and bone density will be assessed radiographically.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from missing single or multiple maxillay anterior and /or premolar with at least 8 mm alveolar ridge height, with 4-6mm alveolar buccolingual (BL) ridge width.
* Patients should be systemically healthy.
* Patients available during follow up periods.

Exclusion Criteria:

* Pregnant females.
* Smokers.
* Poor oral hygiene.
* Vulnerable patients

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
assessment of gain in alveolar ridge width | before surgery and immediately after surgery
  Radiographically

SECONDARY OUTCOMES:
primary implant stability | at the end of surgery
  Implant stability quotient measured by ostell
bone density | before surgery and immediately after surgery
  radiographically

CONTACTS AND LOCATIONS:
Overall Officials: Nevine H. El Din, Professor, Study Director — Faculty of Dentistry, Ain Shams University

IPD SHARING:
Plan to Share IPD: No